CLINICAL TRIAL: NCT00658450
Title: A Randomised Trial to Investigate the Effect of a Rehabilitation Program for Cognitive Deficits in Ugandan Children After Cerebral Malaria.
Brief Title: Rehabilitation Program for Cognitive Deficits in Ugandan Children After Cerebral Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Paul Bangirana, Dr Paul Bangirana, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/HD11/4748U
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Malaria, Cerebral
Keywords: Malaria, Cerebral
MeSH Terms: conditions — Malaria, Cerebral | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive rehabilitation training (Experimental): Children in this arm will the receive the intervention comprising of 16 cognitive rehabilitation training (CRT) exercises for 8 weeks. These exercises will train different cognitive skills including attention, visual spatial processing, logical skills and memory.
  Interventions: Behavioral: Cognitive rehabilitation training
- Treatment as usual (No Intervention): Children in this group will not receive any intervention, they will undergo the usual post discharge treatment for brain injured children at Mulago Hospital (the study site). This is the treatment as usual (TAU) group.

INTERVENTIONS:
Behavioral: Cognitive rehabilitation training — A computerised cognitive training package where children will be required to complete several cognitive tasks. The aim is to strengthen the different cognitive processes during these tasks which in turn may lead to improve cognitive processes.
  Children will complete these tasks in 16 session for 8 weeks.
  Other Names: Intervention group
  Arms: Cognitive rehabilitation training

SUMMARY:
The purpose of this study is to determine whether computerised cognitive rehabilitation training improves cognition in children who have had cerebral malaria.

DETAILED DESCRIPTION:
Cerebral malaria affects several children in sub-Saharan Africa leaving some survivors with cognitive problems especially in attention and memory. There are currently no tested interventions for such deficits resulting from infectious diseases like malaria or other causes. Providing such interventions will go a long way in helping these children achieve their full potential.

ELIGIBILITY:
CM group Inclusion Criteria:

* aged five to 15 years, presenting with asexual forms of P. falciparum malaria on a peripheral blood smear, unarousable coma (not able to localize a painful stimulus) and no other cause for coma (normal CSF).

CM group Exclusion Criteria:

* history of or present meningitis, encephalitis, prior CM, sickle cell disease (SCD), HIV infection, epilepsy, multiple seizures, developmental delay and history of hospitalization for malnutrition.

Healthy control group Inclusion Criteria:

* aged five to 15 years with no other illness at present, within two years of the CM child (for CM children aged 5 and 6 years, the HC's age wont go below 5 and for CM children aged 14 and 15, the HC's age wont go above 15 years).

Healthy control group Exclusion Criteria:

* history of or present bacterial meningitis, encephalitis, CM, SCD, HIV infection, history of hospitalization for malnutrition and any chronic illness for which the patient is currently taking medication.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Improvement in attention scores | 6 months

SECONDARY OUTCOMES:
Improvement in memory, reasoning, planning, behaviour and academic achievement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ibingira, MMED, Study Chair — Chairman, Makerere University Faculty of Medicine Research and Ethics Committee
Locations (1):
- Mulago hospital Acute Care Unit and the Cerebral Malaria Project, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Bangirana P, Idro R, John CC, Boivin MJ. Rehabilitation for cognitive impairments after cerebral malaria in African children: strategies and limitations. Trop Med Int Health. 2006 Sep;11(9):1341-9. doi: 10.1111/j.1365-3156.2006.01685.x. PMID 16930255
- [Background] Boivin MJ, Bangirana P, Byarugaba J, Opoka RO, Idro R, Jurek AM, John CC. Cognitive impairment after cerebral malaria in children: a prospective study. Pediatrics. 2007 Feb;119(2):e360-6. doi: 10.1542/peds.2006-2027. Epub 2007 Jan 15. PMID 17224457